CLINICAL TRIAL: NCT01344382
Title: CRAFT: Helping Parents Initiate and Support Their Adolescent's Treatment
Brief Title: Family Training Program for Parents of Substance Using Adolescents
Acronym: FTP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: Robert J. Meyers PhD & Associates (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5P50DA027841-02 (NIH); P50DA027841 (NIH)
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Substance-Related Disorders; Drug Addiction; Substance Abuse
Keywords: Adolescent; Parent; Substance Abuse; Parent Training; Community Reinforcement and Family Training; CRAFT; Community Reinforcement Approach; Addiction; Family Intervention
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — Atrial Natriuretic Factor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRAFT (Experimental): All parents will be scheduled for 12 individual Community Reinforcement and Family Training for parents (CRAFT-P) training sessions within 120 days and allowed to use up to 6 additional emergency sessions at any time up to the 12-mo follow-up. The first session will last 90 min; the remaining sessions will be 50 - 60 min in duration. Emergency sessions typically last 30 - 60 min and are used to assist the parent with crisis situations during the treatment period (e.g., adolescent violence, arrest) or for booster sessions after.
  Interventions: Behavioral: Community Reinforcement and Family Training
- Al-Anon Facilitation (Active Comparator): All parents will be scheduled for 12 individual Alanon/Naranon Facilitation Training (ANF) sessions within 120 days and allowed to use up to 6 additional emergency sessions at any time up to the 12-mo follow-up. The first session will last 90 min; the remaining sessions will be 50 - 60 min in duration. Emergency sessions typically last 30 - 60 min and are used to assist the parent with crisis situations during the treatment period (e.g., adolescent violence, arrest) or for booster sessions after.
  Interventions: Behavioral: Al-Anon Facilitation

INTERVENTIONS:
Behavioral: Community Reinforcement and Family Training — The philosophy of Community Reinforcement and Family Training (CRAFT) is that drug abuse is caused by multiple biological and environmental factors, many of which are beyond the parents' control. However, because parents have an important relationship with their child, they may able to influence his or her behavior. CRAFT for parents (CRAFT-P) will teach the parent new ways to interact with their child. Sessions will be designed to build the parents' motivation to comply with the training, conduct a functional analysis of their child's drug use pattern, train methods of behavior management and communication skills, enrich the parent's life and to suggest and motivate treatment entry.
  Other Names: CRAFT
  Arms: CRAFT
Behavioral: Al-Anon Facilitation — Al-Anon Facilitation (ANF) parallels the Twelve Step Facilitation intervention developed by Nowinski et al. (1992) for Project MATCH. The content focuses on introducing parents to Alanon or Naranon's purpose and philosophy, educating about 12-step concepts, the fellowship community, denial and enabling, acceptance, caring detachment, and surrendering to a higher power. The trainer's role is to help the parent to gain insight into the ways they interact with their child and to educate and encourage the parent to become actively involved in a 12-step community and to take advantage of its many offerings.
  Other Names: ANF
  Arms: Al-Anon Facilitation

SUMMARY:
This project will modify Community Reinforcement and Family Training (CRAFT; n=15) and Alanon/Naranon Facilitation (ANF; n=15) for use with parents who are concerned about an out-of-treatment adolescent. ANF was selected as a comparison because Alanon and Naranon are the most commonly available method for helping family members. The investigators will compare CRAFT for parents (CRAFT-P) (n=77) and ANF (n=77) to determine if there is a significant difference in adolescent treatment entry. Parents will attend a maximum of 18 sessions with a family specialist and also complete questionnaires periodically over a 12-month period. Parents' adolescents will have the opportunity to participate in the study by completing questionnaires at the same time points as their parent. Our primary hypothesis asks whether participants who are enrolled in the CRAFT-P condition will report more adolescent treatment entry than the ANF condition. Our secondary hypotheses examine: 1) reductions in adolescent substance use and behavior problems in the CRAFT-P group compared to the ANF condition, 2) improvements in parenting skills in the CRAFT-P group compared to the ANF condition and 3) significant pre to post treatment effects for improvements in social functioning, mood, and in parent-adolescent relationship satisfaction.

DETAILED DESCRIPTION:
Data suggest that as many as 60% of parents who are aware and concerned about their adolescent's substance use are unable to get them into treatment without assistance (Szapocznik et al., 1988) and very little research has examined methods to help them. Community Reinforcement and Family Training (CRAFT) was developed to help family members foster treatment entry of treatment-resistant adults, but it has not been tested in a controlled trial with parents of substance-abusing adolescents. This project will modify CRAFT (CRAFT-P) and Alanon/Naranon Facilitation (ANF) for use with parents who are concerned about an out-of-treatment adolescent.

The purpose of this study is to examine the efficacy of the CRAFT-P program in helping parents to: 1) facilitate treatment entry of their child, 2) achieve the outcomes they desire for their adolescents, 3) improve parenting skills in general and in acquisition of CRAFT knowledge in particular, and 4) improve their own mood and functioning. In addition the investigators will examine parents whose child entered treatment to estimate effect sizes of the new CRAFT methods for facilitating parent-supported treatment retention and aftercare engagement in community-based settings. Finally, if the CRAFT program appears efficacious, additional translational work will be initiated in collaboration with the Partnership at Drugfree.org (formerly the Partnership for a Drug-Free America) to provide parents with direct access to components of the CRAFT program.

A Stage II two-group randomized controlled clinical trial will compare CRAFT-P vs ANF. The investigators will collect data from approximately 308 participants (154 parents and 154 adolescents) and each participant will be involved in the study for a maximum of 12 months. The total enrollment number is not exact because it is possible that some adolescents will decline to participate.

Parents will be screened to determine their eligibility. If eligible and interested in participating in the study, the parent will then provide informed consent and give permission for their adolescent to participate in the study. Parents will be randomized to one of the two interventions, CRAFT-P or ANF. Each session will be audio-recorded and stored so that the investigators can complete on-going monitoring to minimize condition bleeding and protect against trainer drift. In addition to completing screening and baseline assessments, parents and adolescents will complete full assessment batteries at 3-, 6-, & 12-months post-baseline. The adolescents' research participation involves completing the assessment battery only and these data will be compared to parent reports to examine consistency.

ELIGIBILITY:
Inclusion Criteria:

Parent Criteria

1. parent is over 21 yrs old
2. parent expresses concern about the drug abuse of their adolescent or young adult
3. parent has the ability to have face-to-face contact with the child on at least 15 out of 30 days with no planned decrease in the amount of contact in the next 12 mo
4. parent has an adolescent or young adult with primary drug abuse of alcohol or a psychoactive drug other than tobacco or caffeine
5. the adolescent/young adult is between 12-25 yrs old at time of consent
6. the child is not receiving treatment addressing the drug abuse/dependence and is not willing for treatment at the time of parental study consent

Adolescent/Young Adult Criteria

1. child's parent meets all eligibility criteria and consents to participate

Exclusion Criteria:

Parent Criteria

1. parent does not agree to participate
2. parent who is providing consent does not demonstrate understanding of participation by reading the consent form and passing a consent quiz testing comprehension of basic elements of informed consent and requirements of the protocol
3. parent is not willing and able to provide valid locator information, to allow training sessions to be recorded, and/or to complete follow-up assessments (determined via consent quiz)
4. parent has a drug abuse problem themselves as determined through PSUD (DSM-IV-TR criteria)
5. parent has a history of drug abuse or dependence and has not been in recovery for more than 2 yrs
6. parent is in a close relationship with another participant such that their participation is unlikely to be independent
7. parent is not able to comprehend the content in the questionnaires even after it is explained several times
8. parent or adolescent/young adult has been diagnosed as having or behaves in a manner consistent with having significant cognitive impairment (e.g., unremitting psychosis, dementia, or other severe psychiatric disorder)
9. parent is currently receiving treatment that addresses the adolescent's substance use (e.g., family therapy)
10. adolescent has a recent history of severe violence toward the parent(s) (e.g., involving weapons, serious injury, or hospitalization).

Adolescent/Young Adult Criteria

1. adolescent/young adult does not agree to participate
2. adolescent/young adult who is providing consent or assent does not demonstrate understanding of participation by reading the consent/assent form and passing a quiz testing comprehension of basic elements of informed consent and requirements of the protocol
3. adolescent/young adult is not able to comprehend the content in the questionnaires even after it is explained several times
4. adolescent/young adult has been diagnosed as having or behaves in a manner consistent with having significant cognitive impairment (e.g., unremitting psychosis, dementia, or other severe psychiatric disorder)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Treatment Entry | Each session and 3-, 6-, and 12-months post-baseline
  The primary outcome measure is treatment entry of the adolescent substance user. This data will be collected via the Supplemental Services Form which is completed by parent participants prior to each session with their specialist and during follow-up assessments. The form is also completed by the adolescent at each follow-up up assessment. Parents or adolescents may also inform study staff of treatment entry at any time during the study.

SECONDARY OUTCOMES:
Adolescent Substance Use | Baseline and 3-, 6-, and 12- months post-baseline
  We will assess adolescent substance use in two ways. Parents will complete the Timeline Follow Back about their adolescent's drug use and the adolescents will also complete the Timeline Follow Back if they're a study participant. In addition, adolescent study participants will give a urine sample to be tested for 8 drugs during each follow-up assessment.
Adolescent Behavior Problems | Baseline and 3-, 6-, and 12-months post baseline
  Adolescent behavior problems will be measured with the Child Behavior Checklist or Adult Behavior Checklist(completed by parent participants) and the Youth Self Report or Adult Self Report(completed by adolescent/Young Adult participants).
Improvement in Parenting Skills | Baseline and 3-, 6-, and 12-months post-baseline
  The Adolescent Parenting Questionnaire will be completed by parent participants. In addition, parents will complete the Family Training Survey and the Parent Role Play Assessment to assess CRAFT knowledge.
Parent Social Functioning | Baseline and 3-, 6-, and 12-months post-baselin
  Social functioning will be measured using the Stress Index for Parents of Adolescents
Parent Mood | Baseline and 3-, 6-, and 12-months post-baseline
  Parent mood will be measured with the Profile of Mood States Questionnaire Brief Form.
Relationship Satisfaction | Baseline and 3-, 6-, 12-months post-baseline
  Parent participants will complete the Parent Happiness with Youth Scale to measure relationship satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly C Kirby, PhD, Principal Investigator — Treatment Research Institute
Locations (1):
- Family Training Program, Philadelphia, Pennsylvania, United States